CLINICAL TRIAL: NCT02956967
Title: Home Administration Of Nivestim(tm) In The Primary Prophylaxis Of Chemotherapy- Induced Febrile Neutropenia Non-interventional, Observational, Prospective Study Short Name: Home Short Name: Home
Brief Title: Home Administration of NivestimTM in the Primary Prophylaxis of Chemotherapy-Induced Febrile Neutropenia
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: ZOB-NIV-1504; C1121004 (Other: Alias Study Number)
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Non-Interventional Study
Keywords: Non-Interventional Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving Nivestim
  Interventions: Other: Overall satisfaction questionnaires of home use of Nivestim

INTERVENTIONS:
Other: Overall satisfaction questionnaires of home use of Nivestim

SUMMARY:
Non-interventional, non-comparative, national, multi-site, single-arm prospective observational study to investigate home administration of Nivestim in the primary prophylaxis of chemotherapy-Induced febrile neutropenia

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years
* Declaration of informed consent signed by patient
* Patients with a solid tumour or with a malignant haematological tumour
* Patients who have been prescribed cytotoxic chemotherapy, irrespective of current cycle
* GCSF-naïve patients or patients pre-treated with GCSF who received no GCSF in the last three months before enrolment
* Patients starting primary prophylactic treatment using NivestimTM either to shorten the duration of a neutropenia or to prevent the occurrence of chemotherapy-induced FN

Exclusion Criteria:

* Patients with chronic myeloid leukaemia (CML) or with myelodysplastic syndrome (MDS)
* Patients who are hypersensitive to one of the excipients of NivestimTM
* Patients not undergoing chemotherapy
* Patients being treated curatively or as secondary prophylaxis with G-CSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing cytotoxic chemotherapy treated prophylactically with NivestimTM in order to reduce the duration of neutropenia and to reduce the incidence of chemotherapy-induced FN.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- Germany (28):
  - Office of Manfred Welslau, Aschaffenburg
  - Office of Martine Klausmann, Aschaffenburg
  - Office of Bernhard Heinrich, Augsburg
  - Campus Charite Mitte, Med. Klinik m. Schwerpunkt Haematologie und Onkologie, Berlin
  - Office of Reinhard Musch, Berlin
  - Office of Peter Klare, Berlin
  - Office of Ute Bückner, Bochum
  - Office of Peter Jungberg, Chemnitz
  - Office of Ivo Azeh, Gelsenkirchen
  - Office of Peter von Wussow, Hanover
  - Office of Volker Petersen, Heidenheim
  - Office of Lars-Jörgen Hahn, Herne
  - Office of Michael Neise, Krefeld
  - Office of Gunther Rogmans, Krefeld
  - Office of Peter Anhut, Kronach
  - Office of Albrecht Kretzschmar, Leipzig
  - Office of Nidal Gazawi, Leipzig
  - Office of Udo Hieber, Mannheim
  - Office of Christoph Salat, München
  - Office of Christian Lerchenmüller, Münster
  - Office of Burkhard Otremba, Oldenburg
  - Office of Julian Topaly, Osnabrück
  - Office of Andre-Robert Rotmann, Rodgau
  - Office of Rene Schubert, Scheibenberg
  - Office of Matthias Groschek, Stolberg
  - Office of Carsten Hielscher, Stralsund
  - Office of Thomas Kuhn, Stuttgart
  - Office of Ortwin Klein, Wiesbaden

REFERENCES:
- [Derived] Otremba B, Hielscher C, Petersen V, Petrik C. Home administration of filgrastim (Nivestim) in primary prophylaxis of chemotherapy-induced febrile neutropenia. Patient Prefer Adherence. 2018 Oct 16;12:2179-2186. doi: 10.2147/PPA.S168029. eCollection 2018. PMID 30410313

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivestim: Participants with an ongoing malignant solid or haematological tumour undergoing cytotoxic chemotherapy and treated prophylactically with subcutaneous Nivestim up to a maximum dose of 48 microgram per day (mcg/day) as per the physician's decision were observed for up to a maximum duration of 6 months in this study. The median duration of treatment cycles was 21 days.
Period: Overall Study
Arm/Group | Nivestim
Started | 171
Completed | 123
Not Completed | 48
Not completed — Adverse Event | 3
Not completed — Reason non-related to neutropenia | 10
Not completed — Lost to Follow-up | 5
Not completed — Missing | 1
Not completed — Termination of Nivestim administration | 29

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants with at least one dose of Nivestim documented in electronic case report form (eCRF).
Groups:
- Nivestim: Participants with an ongoing malignant solid or haematological tumour undergoing cytotoxic chemotherapy and treated prophylactically with subcutaneous Nivestim up to a maximum dose of 48 mcg/day as per the physician's decision were observed for up to a maximum duration of 6 months in this study. The median duration of treatment cycles was 21 days.
Arm/Group | Nivestim
Number analyzed (Participants) | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Significant Comorbidities
Description: Comorbidities included ongoing cardiovascular diseases, liver failure, psychological disorders, respiratory disease, viral infections and other infections (respiratory tract, systemic, uro-genital). Percentage of participants with any ongoing comorbidities were reported in this outcome measure.
Time Frame: Baseline (Day 1)
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF.
Measure: Number; unit: percentage of participants
Arm/Group | Nivestim
Number analyzed (Participants) | 171
percentage of participants | 42.7

2. Primary Outcome: Percentage of Participants With Different Types of Haematological Malignancies
Description: Different types of Haematological malignancies included Hodgkin's lymphoma, leukemia (chronic lymphocytic leukemia), non-Hodgkin's lymphoma and other stem cell transformations. Percentage of participants with different type of ongoing haematological malignancies were reported in this outcome measure.
Time Frame: Baseline (Day 1)
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF.
Measure: Number; unit: percentage of participants
Arm/Group | Nivestim
Number analyzed (Participants) | 171
percentage of participants
  Hodgkin's lymphoma | 0.6
  Leukemia | 1.2
  Non-Hodgkin's lymphoma | 1.8
  Other stem cell transformations | 1.2

3. Primary Outcome: Percentage of Participants With Different Types of Solid Tumour
Description: Different types of solid tumour included tumour of a) Digestive organs such as colon, oesophagus, pancreas, stomach tumour b) Gynaecological organs such as breast, endometrium, ovaries tumour c) Lung organs such as non-small cell lung cancer and small cell lung cancer d) Urological organs such as bladder, prostate gland, testicles tumour e) other organ tumours. Percentage of participants with different types of ongoing solid tumour were reported in this outcome measure.
Time Frame: Baseline (Day 1)
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF.
Measure: Number; unit: percentage of participants
Arm/Group | Nivestim
Number analyzed (Participants) | 171
percentage of participants
  Digestive organ: Colon/Rectum Tumour | 3.5
  Digestive organ: Oesophageal Tumour | 1.2
  Digestive organ: Pancreatic Tumour | 3.5
  Digestive organ: Stomach Tumour | 1.2
  Gynaecological: Breast Tumour | 66.7
  Gynaecological: Endometrial Tumour | 1.2
  Gynaecological: Ovarian Tumour | 4.1
  Lungs: Non-small cell lung cancer | 3.5
  Lungs: Small cell lung cancer | 1.8
  Urological: Bladder Tumour | 0.6
  Urological: Prostate Gland Tumour | 2.9
  Urological: Testicles Tumour | 0.6
  Other organ Tumour | 4.1

4. Primary Outcome: Duration of Solid Tumour in Participants Prior to Enrolment in Study
Description: Time from diagnosis of any previous solid tumour in participants up to the enrolment in the study was recorded at baseline and reported in this outcome measure.
Time Frame: Baseline (Day 1)
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF. Here, N (Number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Nivestim
Number analyzed (Participants) | 163
years | 1.0 (2.86) [0.0 to 1.0]

5. Primary Outcome: Number of Participants Who Received Chemotherapy Prior to Enrolment in Study
Time Frame: Baseline (Day 1)
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF.
Measure: Number; unit: participants
Arm/Group | Nivestim
Number analyzed (Participants) | 171
participants | 51

6. Primary Outcome: Duration of Different Types of Chemotherapies Received by Participants During Study
Time Frame: Baseline up to 6 months
Population: The data for this outcome measure was not collected as it was not planned to be analyzed as prespecified in protocol.
Arm/Group | Nivestim
Number analyzed (Participants) | 0

7. Primary Outcome: Percentage of Participants With Response to Study Treatment
Time Frame: Baseline up to 6 months
Population: The data for this outcome measure was not collected as it was not planned to be analyzed as prespecified in protocol.
Arm/Group | Nivestim
Number analyzed (Participants) | 0

8. Secondary Outcome: Participants' Overall Satisfaction Scores in Response to the Study Treatment
Description: Participants rated the overall satisfaction with Nivestim as part of a questionnaire. The participants were asked to complete the questionnaire at three time points (any 3 time points during the study duration of 6 months). The data from all the three time points was summarized and reported collectively in this outcome measure. The satisfaction was rated on a scale ranging from 1 (minimum score) to 6 (maximum score), where higher scores indicated dissatisfaction with the treatment. For this outcome measure, the within-participant average scores are summarized.
Time Frame: Baseline up to 6 months
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF. Here, N signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nivestim
Number analyzed (Participants) | 167
units on a scale | 1.9 (0.85)

9. Secondary Outcome: Participant's Assessment for Nivestim Packaging
Description: Participants evaluated the packaging of Nivestim as part of a questionnaire. The packaging was rated under the 2 available categories as either easy or complicated. The participants were asked to complete the questionnaire at three time points (any 3 time points during the study duration of 6 months). The data from all the three time points was summarized and reported collectively in this outcome measure. For this outcome measure, the total number of participants in each answer category at at least one of the time points is displayed, that is participants who provided different ratings at the individual time points are included in more than one answer category in this summary.
Time Frame: Baseline up to 6 months
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Nivestim
Number analyzed (Participants) | 169
participants
  Easy | 144
  Complicated | 4
  Missing | 21

10. Secondary Outcome: Participant's Assessment of Injection Site Pain and Tolerability
Description: Participants evaluated the injection site pain and the injection site tolerability of the treatment as part of a questionnaire. The injection site pain was rated under the 5 available categories as: Did not feel anything, did not feel much, light stitch, painful and very painful. Injection site tolerability was also rated under the 5 available categories as: Very good, good, satisfactory, did not tolerate well, did not tolerate at all.The participants were asked to complete the questionnaire at three time points (any 3 time points during the study duration of 6 months). The data from all the three time points was summarized and reported collectively in this outcome measure. For both the injection site pain and tolerability, the total number of participants in each answer category at at least one of the time points is displayed, that is participants who provided different ratings at the individual time points are included in more than one answer category for each of them.
Time Frame: Baseline up to 6 months
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Nivestim
Number analyzed (Participants) | 169
participants
  Injection Site Pain: Did not feel anything | 53
  Injection Site Pain: Did not feel much | 128
  Injection Site Pain: Light stitch | 42
  Injection Site Pain: Painful | 4
  Injection Site Pain: Very painful | 0
  Tolerability: Very good | 107
  Tolerability: Good | 106
  Tolerability: Satisfactory | 12
  Tolerability: Did not tolerate well | 4
  Tolerability: Did not tolerate at all | 0

11. Secondary Outcome: Participant's Assessment of Overall Tolerability of Subcutaneous Injection
Description: Participants evaluated the overall tolerability of subcutaneous injection of treatment as part of a questionnaire. The tolerability was rated under the 5 categories as: Very good, good, satisfactory, did not tolerate well, did not tolerate at all. The participants were asked to complete the questionnaire at three time points (any 3 time points during the study duration of 6 months). The data from all the three time points was summarized and reported collectively in this outcome measure. For this outcome measure, the total number of participants in each answer category at at least one of the time points is displayed, that is participants who provided different ratings at the individual time points are included in more than one answer category in this summary.
Time Frame: Baseline up to 6 months
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Nivestim
Number analyzed (Participants) | 169
participants
  Very good | 75
  Good | 117
  Satisfactory | 20
  Did not tolerate well | 14
  Did not tolerate at all | 3

12. Secondary Outcome: Percentage of Participants With Neutropenia
Description: Percentage of participants with absolute neutrophil count (greater than)>0.5*10^9 Neutrophils per Liter were reported in this outcome measure.
Time Frame: Baseline up to 6 months
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF.
Measure: Number; unit: percentage of participants
Arm/Group | Nivestim
Number analyzed (Participants) | 171
percentage of participants | 0.0

13. Secondary Outcome: Percentage of Participants With at Least One Infection and Serious Infection
Description: Infections included bronchitis, upper respiratory tract infection, cystitis, herpes virus infection, influenza, lung infection, oral candidiasis, skin infection and vulvovaginal mycotic infection. Serious Infections included serious adverse events resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 6 months
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF.
Measure: Number; unit: percentage of participants
Arm/Group | Nivestim
Number analyzed (Participants) | 171
percentage of participants
  Infection | 8.2
  Serious Infection | 1.8

14. Secondary Outcome: Change From Baseline in Absolute Neutrophil Count at Cycle 1, 2, 3, 4, 5 and 6
Time Frame: Baseline, Cycle 1, 2, 3, 4, 5, 6
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF. Here, number analyzed (n) signifies those participants who were evaluable at specified time points only.
Measure: Mean (Standard Deviation); unit: 10^9 Neutrophils per Liter
Arm/Group | Nivestim
Number analyzed (Participants) | 171
10^9 Neutrophils per Liter
  Baseline: number analyzed (Participants) | 118
  Baseline | 3.36 (3.005)
  Change at Cycle 1: number analyzed (Participants) | 86
  Change at Cycle 1 | -0.03 (0.528)
  Change at Cycle 2: number analyzed (Participants) | 92
  Change at Cycle 2 | 1.76 (5.304)
  Change at Cycle 3: number analyzed (Participants) | 85
  Change at Cycle 3 | 1.35 (4.787)
  Change at Cycle 4: number analyzed (Participants) | 7
  Change at Cycle 4 | 3.49 (1.924)
  Change at Cycle 5: number analyzed (Participants) | 3
  Change at Cycle 5 | 4.50 (4.107)
  Change at Cycle 6: number analyzed (Participants) | 2
  Change at Cycle 6 | 1.00 (1.556)

15. Secondary Outcome: Minimum Value of Absolute Neutrophil Count
Time Frame: Cycle 1, 2, 3, 4, 5, 6
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF. Here, n signifies those participants who were evaluable at specified time points only.
Measure: Mean (Standard Deviation); unit: 10^9 Neutrophils per Liter
Arm/Group | Nivestim
Number analyzed (Participants) | 171
10^9 Neutrophils per Liter
  Cycle 1: number analyzed (Participants) | 89
  Cycle 1 | 2.49 (3.271)
  Cycle 2: number analyzed (Participants) | 65
  Cycle 2 | 3.12 (3.485)
  Cycle 3: number analyzed (Participants) | 66
  Cycle 3 | 2.95 (3.015)
  Cycle 4: number analyzed (Participants) | 4
  Cycle 4 | 4.90 (1.941)
  Cycle 5: number analyzed (Participants) | 1
  Cycle 5 | 9.20 (NA) — As only 1 participant was analyzed at Cycle 5, standard deviation could not be calculated.
  Cycle 6: number analyzed (Participants) | 2
  Cycle 6 | 4.15 (0.354)

16. Secondary Outcome: Absolute Neutrophil Count at the Last Visit During Each Treatment Cycle
Time Frame: End of study visit of Cycle 1, 2, 3, 4, 5, 6 (maximum up to Month 6)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: 10^9 Neutrophils per Liter
Arm/Group | Nivestim
Number analyzed (Participants) | 171
10^9 Neutrophils per Liter
  Cycle 1: number analyzed (Participants) | 71
  Cycle 1 | 8.22 (9.874)
  Cycle 2: number analyzed (Participants) | 62
  Cycle 2 | 6.50 (6.297)
  Cycle 3: number analyzed (Participants) | 65
  Cycle 3 | 6.52 (7.570)
  Cycle 4: number analyzed (Participants) | 4
  Cycle 4 | 1.78 (0.873)
  Cycle 5: number analyzed (Participants) | 1
  Cycle 5 | 0.70 (NA) — As only 1 participant was analyzed at Cycle 5, standard deviation could not be calculated.
  Cycle 6: number analyzed (Participants) | 2
  Cycle 6 | 46.15 (51.831)

17. Secondary Outcome: Difference Between Minimum Value of Absolute Neutrophil Count and Absolute Neutrophil Count
Time Frame: Cycle 1, 2, 3, 4, 5, 6
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: 10^9 Neutrophils per Liter
Arm/Group | Nivestim
Number analyzed (Participants) | 171
10^9 Neutrophils per Liter
  Cycle 1: number analyzed (Participants) | 66
  Cycle 1 | 6.18 (9.548)
  Cycle 2: number analyzed (Participants) | 58
  Cycle 2 | 3.26 (5.872)
  Cycle 3: number analyzed (Participants) | 59
  Cycle 3 | 3.70 (7.450)
  Cycle 4: number analyzed (Participants) | 4
  Cycle 4 | -3.13 (2.653)
  Cycle 5: number analyzed (Participants) | 1
  Cycle 5 | -8.50 (NA) — As only 1 participant was analyzed at Cycle 5, standard deviation could not be calculated.
  Cycle 6: number analyzed (Participants) | 2
  Cycle 6 | 42.00 (52.184)

18. Secondary Outcome: Duration From Minimum Value of Absolute Neutrophil Count to the Absolute Neutrophil Count
Time Frame: Cycle 1, 2, 3, 4, 5, 6
Population: as for outcome 15
Measure: Median (Full Range); unit: days
Arm/Group | Nivestim
Number analyzed (Participants) | 171
days
  Cycle 1: number analyzed (Participants) | 90
  Cycle 1 | 5.0 [-9 to 28]
  Cycle 2: number analyzed (Participants) | 65
  Cycle 2 | 4.0 [-17 to 41]
  Cycle 3: number analyzed (Participants) | 69
  Cycle 3 | 4.0 [-9 to 18]
  Cycle 4: number analyzed (Participants) | 3
  Cycle 4 | 6.0 [5 to 7]
  Cycle 5: number analyzed (Participants) | 1
  Cycle 5 | 9.0 [9.0 to 9.0]
  Cycle 6: number analyzed (Participants) | 2
  Cycle 6 | 5.5 [5.0 to 6.0]

19. Secondary Outcome: Percentage of Participants With Febrile Neutropenia
Description: Grade 3/4 febrile neutropenia is defined as a temperature of greater than or equal to (>=) 38.0 degree Celsius and absolute neutrophil count of less than (<) 1.0 × 10^9 Neutrophils per Liter.
Time Frame: Baseline up to 6 months
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF.
Measure: Number; unit: percentage of participants
Arm/Group | Nivestim
Number analyzed (Participants) | 171
percentage of participants | 0.6

20. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; cancer; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 6 months that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious.
Time Frame: Baseline up to 6 months
Population: Full analysis set included all participants with at least one dose of Nivestim documented in eCRF.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivestim
Number analyzed (Participants) | 171
Participants
  AEs | 81
  SAEs | 16

ADVERSE EVENTS:
Time Frame: Baseline up to 6 months
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Nivestim
All-Cause Mortality (participants affected / at risk) | 0/171
Serious Adverse Events (participants affected / at risk) | 16/171
Other Adverse Events (participants affected / at risk) | 74/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivestim (N=171)
Chest pain (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Pain (General disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
General physical health deterioration (General disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Athralgia (Musculoskeletal and connective tissue disorders) | 1
Infection (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivestim (N=171)
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Pyrexia (General disorders) | 4
Fatigue (General disorders) | 3
Mucosal Inflammation (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 3
Asthenia (General disorders) | 2
Chills (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site erythema (General disorders) | 1
Malaise (General disorders) | 1
Mucosal toxicity (General disorders) | 1
Peripheral swelling (General disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 8
Anaemia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Cytopenia (Blood and lymphatic system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Dysaesthesia (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Bronchitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Platelet count increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Tachycardia (Cardiac disorders) | 2
Cardiovascular disorder (Cardiac disorders) | 1
Cardiovascular insufficiency (Cardiac disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Axillary vein thrombosis (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Blepharospasm (Eye disorders) | 1
Visual Impairment (Eye disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.